CLINICAL TRIAL: NCT02203942
Title: Comparing NAAT Testing to Standard Methods in Diagnosis of Vaginal Infections in the General Gynecology and Vulvovaginal Referral Offices.
Brief Title: Comparing NAAT Testing to Standard Methods for the Diagnosis of Vaginitis
Acronym: VAST
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Harold Wiesenfeld, Associate Professor, University of Pittsburgh
Other Study IDs: PRO14010349
Record Dates: First submitted 2014-07-25; First posted 2014-07-30 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Bacterial Vaginosis; Vulvovaginal Candidiasis; Trichomoniasis
Keywords: Bacterial Vaginosis; Vulvovaginal Candidiasis; Trichomoniasis
MeSH Terms: conditions — Vaginosis, Bacterial; Candidiasis, Vulvovaginal; Trichomonas Infections

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vaginal Infections (BV, VVC, trich): NAAT testing Amsel criteria Nugent score yeast culture TV culture
  Interventions: Other: NAAT testing

INTERVENTIONS:
Other: NAAT testing — comparison of NAAT testing for BV, VVC and trich to Amsel criteria, Nugent score, yeast culture and TV culture.

SUMMARY:
Vaginitis is the most common condition encountered in the gynecologist's office and is most commonly caused by bacerial vaginosis (BV), vulvovaginal candidiasis (VVC) and Trichomonas vaginalis (TV). Establishing the correct etiology of symptomatic vaginitis can be challenging, and the evaluation of vaginitis by physicians is often substandard.

The investigators will determine whether NAAT testing will improve the diagnosis of vaginal infections including bacterial vaginosis (BV), vulvovaginal candidiasis (VVC) and Trichomonas vaginalis (TV).

DETAILED DESCRIPTION:
Several commercial nucleic acid amplification tests (NAAT) are available to identify causative organisms. One of these commercial tests has undergone validation published in a scientific journal, only in an STD clinic population. The primary outcome of this study is to compare NAAT diagnostic methods to traditional gold-standard tests for BV, VVC and TV in symptomatic and asymptomatic women in the general gynecology office as well as in a vulvovaginitis referral office. Addressing incorrect evaluation and diagnosis will lead to correct treatment for women suffering from vaginitis.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants aged 18 and older
2. Based on symptoms:

   * Symptomatic patients: with symptoms of vaginitis that include abnormal discharge, malodor, itching, irritation and / or discomfort
   * Asymptomatic controls: no vulvovaginal symptoms
3. Willing to provide written informed consent for participation in this study

Exclusion Criteria:

1. Use of oral antibiotics in the past 14 days
2. Use of vaginal products or lubricant, vaginal intercourse, or douching in the last 24 hour

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Enrollments will include patients seeking care at Magee-Womens Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Vaginal Infections | approximately 7 days
  Compare the sensitivity and specificity of NAAT tests to Amsel criteria, Nugent score for bacterial vaginosis, yeast culture and TV culture in detecting BV, VVC, and trichomoniasis.

CONTACTS AND LOCATIONS:
Overall Officials: Harold C Wiesenfeld, MD, CM, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States